CLINICAL TRIAL: NCT07001982
Title: The Relationship Central Sensitization, Pain and Depression Patients With Lumbar Spinal Stenosis
Brief Title: Lumbar Spinal Stenosis and Central Sensitization
Status: Recruiting | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Musa Güneş, Principal Investigator, PhD, Karabuk University
Other Study IDs: Karabuk-2325
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with central sensitization with LSS: Patients with lumbar spinal stenosis with high sensitization will be included.
- Normal sensitization patients with LSS: Patients with lumbar spinal stenosis with normal sensitization will be included.

SUMMARY:
Lumbar spinal stenosis (LSS) functionally limits individuals by causing pain in both the waist and the legs during activity and walking. Pain is, therefore, an important problem for patients. Pain lasts for years in LSS and thus becomes chronically persistent. As a result, persistent pain can cause sensitization due to a decrease in the pain threshold. This condition affects patients not only biomedically but also biopsychosocially. For this reason, various sleep disorders and mood disorders can develop in patients. Therefore, this study aimed to examine the relationship between central sensitization and pain, disability, sleep and depression in patients with LSS.

DETAILED DESCRIPTION:
Lumbar spinal stenosis (LSS) functionally limits individuals by causing pain in both the waist and the legs during activity and walking. In particular, the pain in LSS lasts for years and becomes chronic and can cause persistent and disturbing sensitization. This situation may be associated with decreased pain threshold and allodynia. Various studies show that sensitization can affect individuals biomedically and may lead to important health problems. Some of these are sleep and depression problems. Sleep and a healthy mentality are important for continuing daily activities and preserving quality of life. However, when the literature is examined, it is seen that central sensitization and the parameters that may be related to this have not been examined sufficiently. Therefore, the aim of this study is to examine the relationship between central sensitization and pain, disability, sleep and depression in patients with LSS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with lumbar spinal stenosis by MRI,
* The ages of 45-80,
* Low back and/or leg pain that has persisted for at least 3 months
* Volunteer to participate in the study

Exclusion Criteria:

* Patients who did not agree to participate in the study,
* Those with a history of serious neurological diseases such as Parkinson's, hemiplegia, multiple sclerosis,
* Those who had undergone surgery in the lumbar region within the last year,
* Those with advanced joint disease in the lower extremity,
* Those with malignancy in the spine,
* Those who had a previous operation for the lower extremity,
* Those who had a pain or disability in other musculoskeletal joints,
* Those who had a psychological disorder or peripheral vascular disease
* Those who had any concurrent serious medical condition, including sepsis or cancer
* Those who did not cooperate well were not included in the study.

Ages: 45 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with lumbar spinal stenosis will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Central sensitization | Baseline
  Central sensitization will be assessed with the "Central Sensitization Scale". The total score range is between 0-100 points. As the score increases, sensitization increases and 40 points and above are considered higher sensitization.
Pain severity | Baseline
  Pain intensity will be assessed with Numeric Rating Scale (NRS). NRS varies between 0-10 and the higher the score, the greater the pain.
Pain pressure threshold | Baseline
  Pressure pain threshold will be measured with an algometer in kg. High values indicate a high pain threshold.
Disability levels | Baseline
  Disability will be measured by the Oswestry Disability Index. The total score ranges from 0-100 and the higher the score, the higher the level of disability.
Pain catastrophizing | Baseline
  It will be evaluated using the pain catastrophizing scale. The total score varies between 0-52. As the score increases, negative feelings and thoughts increase.
Sleep quality | Baseline
  Sleep quality will be assessed with the Pittsburgh Sleep Quality Index. It is scored from 0 to 21, with higher scores indicating worse sleep quality.
Depression | Baseline
  The Center for Epidemiological Studies Depression Scale (CES-D) will be used to assess depression.The total score is 0-60. As the score increases, depression increases.

CONTACTS AND LOCATIONS:
Overall Officials: Musa Güneş, PhD, Study Director — Karabuk University
Locations (1):
- Karabuk University, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Iwasaki R, Miki T, Miyazaki M, Kanetaka C, Mitsuyama T, Ota K. Neuropathic Pain Was Associated with Central Sensitivity Syndrome in Patients with Preoperative Lumbar Spinal Stenosis Using the painDETECT and Central Sensitization Inventory Questionnaires: A Cross-Sectional Study. Pain Res Manag. 2023 May 10;2023:9963627. doi: 10.1155/2023/9963627. eCollection 2023. PMID 37207128
- [Result] Ogon I, Takashima H, Morita T, Fukushi R, Takebayashi T, Teramoto A. Association of central sensitization, visceral fat, and surgical outcomes in lumbar spinal stenosis. J Orthop Surg Res. 2023 Nov 21;18(1):886. doi: 10.1186/s13018-023-04376-2. PMID 37990264